CLINICAL TRIAL: NCT05072964
Title: The FARAPULSE FARA-Freedom Trial A Prospective Open Label Single Arm Post Market Clinical Follow-Up Trial of the FARAPULSE Pulsed Field Ablation System in Patients With Paroxysmal Atrial Fibrillation
Brief Title: The FARAPULSE FARA-Freedom Trial
Acronym: FARA-Freedom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1169
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Catheter Ablation; Pulmonary Vein Isolation (PVI); Atrial Fibrillation (AF); Atrial Flutter; Atrial Tachycardia; Pulsed Field Ablation; Cavo-tricuspid isthmus; Anti-arrhythmic drugs; Atrial Fibrillation Drugs; Cardiac Arrhythmias; Cardiac Ablation; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE Pulsed Field Ablation System (Other): Ablation using the FARAPULSE Pulsed Field Ablation System
  Interventions: Device: FARAPULSE Pulsed Field Ablation System

INTERVENTIONS:
Device: FARAPULSE Pulsed Field Ablation System — A pulmonary vein isolation will be performed using catheter ablation
  Other Names: Ablation catheters indicated for Paroxysmal Atrial Fibrillation

SUMMARY:
The Post-Market Clinical Follow-Up trial is a prospective, multi-center, open-label, single-arm clinical follow-up study designed to provide long-term safety feasibility, effectiveness and performance of the FARAPULSE Pulsed Field Ablation System for the treatment of Paroxysmal Atrial Fibrillation (PAF).

DETAILED DESCRIPTION:
The primary and secondary Safety, Feasibility, Effectiveness and Performance will be evaluated against pre-specified criteria as determined by the Sponsor and FDA. The criteria set in this study have been previously used to demonstrate Safety, Feasibility, Effectiveness and Performance in FARAPULSE Pulsed Field Ablation System for the treatment of Paroxysmal Atrial Fibrillation (PAF).

The analysis of the primary safety and performance objective will take place once all the subjects with a study FARAPULSE Pulsed field ablation procedure attempt have reached 12 months of follow-up post-pulsed field ablation procedure.

The analyses of the primary effectiveness objective will take place once all the subjects with a study pulsed field ablation procedure attempt have reached 34 ~ 36 months of follow-up post-pulsed field ablation procedure.

The analyses for the secondary objectives will take place once all subjects with a study pulsed field ablation procedure attempt have reached 34~36 months of follow-up post-pulsed field ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paroxysmal atrial fibrillation (PAF), AND
* Two (2) or more episodes of recurrent PAF during the 6 months preceding the consent Date, AND
* At least 1 episode of Atrial Fibrillation (AF) documented with a tracing within 12 months preceding the consent date.
* Age 18 years or older
* Therapeutic Failure for the treatment of Atrial Fibrillation (effectiveness or intolerance) of at least one active antiarrhythmic drug (AAD) for rhythm control.
* Willing and Capable of providing Informed Consent to undergo study procedures AND
* Participate in all examinations and follow-up visits and tests associated with this clinical study

Exclusion Criteria:

* Any previous left atrial (LA) ablation (except permissible retreatment subjects)
* Any previous LA surgery
* Current intracardiac thrombus (can be treated after thrombus is resolved)
* Presence of any pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Body Mass Index (BMI) >45.0
* Anteroposterior Left Atrial diameter > 5.5 cm by transthoracic echocardiography (TTE)/ intracardiac imaging (ICE)
* Presence of any cardiac valve prosthesis
* Clinically significant mitral valve regurgitation or stenosis
* Myocardial infarction, percutaneous coronary intervention (PCI) / percutaneous transluminal coronary angiography (PTCA) or coronary artery stenting which occurred during the 3 month interval preceding the Consent Date
* Unstable angina
* Any cardiac surgery which occurred during the 3 month interval preceding the Consent Date
* Any significant congenital heart defect corrected or not (including atrial septal defects or pulmonary vein abnormalities but not including minor PFO)
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) < 35%
* 2º (Type II) or 3º atrioventricular block
* Presence of a permanent pacemaker, biventricular pacemaker, atrial defibrillator or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
* Hypertrophic cardiomyopathy
* Active Systemic infection
* Uncontrolled hyperthyroidism
* Any cerebral ischemic event (strokes or TIAs) which occurred during the 6 month interval preceding the Consent Date.
* Any woman known to be pregnant
* Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
* Severe lung disease, pulmonary hypertension, or any lung disease associated with chronic abnormal blood gases or requiring supplemental oxygen
* Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
* Active malignancy, or history of treated malignancy within 24 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma)
* Life expectancy less than one (1) year
* Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study (data collection for registries or retrospective studies is permitted)
* Unwilling or unable to comply fully with study procedures and follow-up
* Clinically significant psychological condition that in the Investigator's opinion would prohibit the subject's ability to meet the protocol requirements
* Other uncontrolled medical conditions that may modify device effect or increase risk, including uncontrolled diabetes mellitus, untreated sleep apnea or active alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (2):
  - AZ Sint-Jan Brugee, Bruges
  - Jessa Ziekenhuis, Hasselt
- Czechia (3):
  - Neuron Medical, Brno
  - Nemocnice Na Homolce, Prague
  - IKEM Cardiac Center, Prague
- Copenhagen(Gentofte) Hospital, Hellerup, Denmark
- Germany (4):
  - Heart- and Diabetescenter NRW, Bad Oeynhausen
  - CCB Frankfurt, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios-Hamburg,Germany, Hamburg
- Netherlands (2):
  - Catherina, Eindhoven
  - UMCG, Groningen
- Inselspital - Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzner A, Fiala M, Vijgen J, Ouss A, Gunawardene M, Hansen J, Kautzner J, Schmidt B, Duytschaever M, Reichlin T, Blaauw Y, Sommer P, Vanderper A, Achyutha AB, Johnson M, Raybuck JD, Neuzil P. Long-term outcomes of the pentaspline pulsed-field ablation catheter for the treatment of paroxysmal atrial fibrillation: results of the prospective, multicentre FARA-Freedom Study. Europace. 2024 Mar 1;26(3):euae053. doi: 10.1093/europace/euae053. PMID 38385529

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE Pulsed Field Ablation System
Started | 180
Completed | 175
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 18
  Belgium | 28
  Czechia | 63
  Denmark | 12
  Switzerland | 9
  Germany | 50

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Percentage of Participants Free of Chronic Treatment Failure Through 12 Months and Freedom From Recurrence of Symptomatic Atrial Fibrillation, Atrial Tachycardia or Atrial Flutter
Description: Evaluated by assessing the rate of subjects free of chronic treatment failure with paroxysmal atrial fibrillation who have failed one Antiarrhythmic Drugs (AAD).
  Includes both acute procedural success ( Demonstration of Acute Vein Success in all attempted PVs using the FARAPULSE Pulsed Field Ablation System during the first ablation procedure (Index or or rescheduled index Procedure
Time Frame: 12 Months
Population: Modified Intent To Treat
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 180
Participants | 121

2. Primary Outcome: Safety: Percentage of Participants Experiencing Composite Safety Endpoint(CSE) Through 12 Months
Description: To demonstrate safety of FARAPULSE Pulsed Field Ablation System, by assessing the rate of subjects experiencing Early and Late onset Composite Safety Endpoints(CSE) with paroxysmal atrial fibrillation who have therapeutic failure of at least one AntiArrhythmic Drug (AAD)
Time Frame: 12 Months
Population: Modified Intent To Treat
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 180
Participants | 2

3. Secondary Outcome: Additional Safety Analyses: Percentage of Participants Free From Any of the Device or Procedure Related SAE
Description: Freedom from a serious adverse event (SAE) which has not been categorized as a Pulsed Field Ablation procedure event.
Time Frame: 12 Months
Population: Modified Intent To treat
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 180
Participants
  Participants free from any of the procedure related SAE | 173
  Participants free from any of the device related SAE | 179

4. Secondary Outcome: Additional Performance Analyses: Acute Procedural Success
Description: Acute Procedural success is the demonstration of Acute Vein Success (measured by % subjects) was determined by Isolation of an ablated PVI using the FARAPULSE Pulsed Field Ablation System during the first ablation procedure (Index or Rescheduled Index Procedure), as clinically assessed by entrance block demonstrated ≥ 20 minutes after the last PVI lesion is made with or without adenosine testing
Time Frame: 1 day
Population: Modified Intent To Treat
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 180
Participants | 180

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE Pulsed Field Ablation System
All-Cause Mortality (participants affected / at risk) | 1/180
Serious Adverse Events (participants affected / at risk) | 25/180
Other Adverse Events (participants affected / at risk) | 9/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=180)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 5 (9)
Atrial Flutter (Cardiac disorders) | 1 (3)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Vascular Psuedoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=180)
Atrial Fibrillation (Cardiac disorders) | 9 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT05072964/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05072964/SAP_001.pdf